CLINICAL TRIAL: NCT04853095
Title: Prospective Randomized Trial Evaluating the Effect of Peritoneal Flap Fixation on Symptomatic and Radiologic Lymphocele Formation Following Robot Assisted Radical Prostatectomy With Extended Pelvic Lymph Node Dissection (PerFix)
Brief Title: Effect of Peritoneal Fixation on Lymphocele Formation
Acronym: PerFix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Olomouc (Other)
Responsible Party: Principal Investigator, Vladimir Student, M.D., Ph.D., Vladimir Student Jr., MD, PhD, FEBU, University Hospital Olomouc
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FNOl 00098892
Record Dates: First submitted 2021-02-28; First posted 2021-04-21 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Prostate Cancer; Lymphocele After Surgical Procedure
Keywords: Prostate cancer; Robot-assisted radical prostatectomy; Extended pelvic lymph node dissection; Lymphocele; Peritoneal fixation; Lymphatic disease
MeSH Terms: conditions — Prostatic Neoplasms; Lymphocele; Lymphatic Diseases | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (PerFix) (Experimental): Peritoneal fixation technique
  Interventions: Procedure: Peritoneal fixation (PerFix)
- Control group (no PerFix) (Active Comparator): Standard of care (i.e. no fixation)
  Interventions: Procedure: Standard of care

INTERVENTIONS:
Procedure: Peritoneal fixation (PerFix) — PerFix involves suturing the free end of the peritoneal flap left after RARP + ePLND to the pelvic wall near the symphysis of the pubic bones leaving two lateral openings for directing the lymphatic fluid out of the pelvis to the abdominal cavity.
  Arms: Intervention group (PerFix)
Procedure: Standard of care — ePLND without peritoneal flap fixation
  Arms: Control group (no PerFix)

SUMMARY:
The PerFix Trial aims to compare the use of peritoneal fixation technique to standard of care (no fixation) during robot-assisted radical prostatectomy with extended pelvic lymph node dissection (RARP + eLND) for the prevention of symptomatic and radiologic lymphocele formation.

DETAILED DESCRIPTION:
Extended pelvic lymph node dissection (ePLND) is the most accurate staging tool to determine lymph node involvement in prostate cancer. As urologist perform this procedure more often now, thanks to the shift to more advanced and aggressive stages, the role of ePLND is expanding. The main complication of PLND is development of a collection of lymphatic fluid called a lymphocele. Lymphoceles can be associated with abdominal pain, lower urinary tract symptoms, bladder outlet obstruction, penile or scrotal edema, infection/sepsis, lower extremity swelling and deep vein thrombosis. They necessitate intervention in up to 10% of patients treated with RARP + ePLND which includes drainage or surgery. Radiologic incidence can be as high as around 50% of operated patients with unknown clinical relevance. Many interventions aimed at reducing the rate of lymphocele formation with limited success so far. Several retrospective studies suggested using peritoneal flap fixation technique which could direct the lymphatic fluid to the peritoneal cavity out of the pelvis and its ensure its reabsorption there. We hypothesize that peritoneal fixation can potentially lower the incidence of symptomatic and radiologic lymphocele formation. By preventing this potentially very dangerous complication, it could be very beneficial for a large group of patients suffering from aggressive localized prostate cancer who are scheduled for RARP + ePLND.

Our goal is to is to test this hypothesis in a randomized trial comparing the fixation technique to standard of care, i.e. no fixation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Able to give informed consent
* Histologically proven high risk prostate cancer or intermediate risk cancer (≥5% risk of nodal involvement on Briganti 2012 nomogram) according to European Association od Urology (EAU) risk groups
* Suitable for minimally-invasive surgery

Exclusion Criteria:

* Previous pelvic surgery or irradiation.
* Any type of clotting disorder.
* Patients unwilling to undergo CT scan
* Kidney failure, Hemodialysis
* American Society of Anesthesiology Classification> 3
* Existing contraindications for performing a lymph node dissection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with Symptomatic lymphocele | 3 months
  The number of participants with symptomatic lymphocele will be determined. Clinical symptoms, time of onset, the size of the lymphocele, location, number of Lymphoceles and intervention needed will be measured

SECONDARY OUTCOMES:
Number of participants with Radiologic lymphocele on pelvic CT scan | 3 months
  The number of participants with radiologic lymphocele on Pelvic CT scan will be determined together with the size, location and number of detected lymphoceles.
Rate of severe (Clavien grade ≥3) complications | 3 months
  Incidence of adverse events in the Prefix group compared to control group (no PerFix) will be measured. Surgical complications will be evaluated according to Clavien-Dindo classification
Change in lymphocele size | 1 year
  The change in lymphocele size during follow-up CT scan will be examined
Number of participants with Occurrence of Any Venous Thromboembolism | 6 months
  Radiologic investigation will be done in case of by swelling or pain of the lower extremity and the number of any venous thromboembolism will be determined
Perioperative outcomes | 30 days
  Perioperative outcomes (time of the surgery, blood loss and hospital stay) will be measured
The effect of lymphocele on urinary incontinence | 1 year
  The rate of continent patients will be defined using pads needed per day. Continent equals to 0-1 pad per day.
The effect of lymphocele on potency | 1 year
  Potency equals to 19 and more points in the International index of erectile function (IIEF5) questionnaire (scale 0-25), the higher the score, the better.
The effect of lymphocele on lower urinary tract symptoms (LUTS) | 1 year
  Change in the International prostate symptom score (IPSS) questionnaire from the baseline will be assessed (scale 0-35, higher score means worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Student, MD, PhD, Principal Investigator — Dpt. of Urology
Locations (1):
- University hospital Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: No